CLINICAL TRIAL: NCT06148168
Title: Comparative Evaluation of Different Doses of Magnesium Sulphate in Oblique Subcostal TAP Block for Laparoscopic Cholecystectomy: a Randomized Double-blind Controlled Study
Brief Title: Magnesium Sulphate in Oblique Subcostal TAP Block
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Yamany Mohamed Kamel, Principle Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Post operative pain
Record Dates: First submitted 2023-10-27; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): 24 patients will receive OSCTAP block with 25 ml volume on each side (5 ml normal saline plus 20 ml of 0.25 % bupivacaine)
  Interventions: Drug: Bupivacaine plus normal saline
- Group B (Active Comparator): 24 patients will receive OSCTAP block with 25 ml volume on each side (5 ml normal saline containing 500 mg MgSO4 plus 20 ml of 0.25% bupivacaine)
  Interventions: Drug: Bupivacaine plus normal saline containing MgSO4
- Group C (Active Comparator): 24 patients will receive OSCTAP block with 25 ml volume on each side (5 ml normal saline containing 250 mg MgSO4 plus 20 ml of 0.25% bupivacain)
  Interventions: Drug: Bupivacaine plus normal saline containing MgSO4

INTERVENTIONS:
Drug: Bupivacaine plus normal saline — Unlike specific peripheral nerve blocks, TAP block is a non-dermatomal "field block". Even with the same US-guided technique, the extent of spread of local anesthetics can be variable due to individual anatomical variations (18). In order to perform the blocks, abdominal skin will be prepared and covered with sterile drapes. The needle can be introduced by multiple punctures along the oblique subcostal line from the xiphoid process towards the anterior part of the iliac crest .Thus, LA will be injected in the TAP along this line provides both upper and lower abdominal wall analgesia. The OSCTAP block more consistently covers L1 dermatome. After negative aspiration, a test injection with 1 ml of 0.9% normal saline will be performed to confirm the needle location. If the intended sensation will not decreased in surgical dermatomes after 30 min, the patient will be regarded to have a failed block and will be excluded from the study.
  Arms: Group A
Drug: Bupivacaine plus normal saline containing MgSO4 — Bupivacaine plus normal saline containing MgSO4
  Arms: Group B; Group C

SUMMARY:
The aim of this study is to evaluate the effect of adding different doses of MgSO4 to bupivacaine via OSCTAB block on postoperative pain control for 24 hours in patients scheduled for LC.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is a gold standard for management of gallbladder stones. Early and easily recovery, less operative morbidities, less postoperative pain, improved cosmetics, less hospitalization days and decreased cost are the superiorities of laparoscopic cholecystectomies over open surgical procedures.

Postoperative pain is the major obstacle for early postoperative ambulation and prolongs the hospital stay. Moreover, it has been hypothesized that intense acute pain after LC may predict development of chronic pain (e.g., post laparoscopic cholecystectomy syndrome). So, aggressive perioperative pain prevention is mandatory.

This pain is routinely managed using opiates, which has several side effects. Transversus abdominis plane (TAP) block is a regional anesthetic technique that has gradually become an alternative for postoperative pain control during laparoscopic abdominal surgeries. It involves the infusion of local anesthetic into the fascial plane of the abdominal wall. Oblique subcostal transversus abdominis plane (OSCTAP) block is an US-guided regional anesthesia technique that anesthetizes the nerves of the lower and upper anterior abdominal wall, specifically from T6 to L1.

Rafi et al and McDonnell et al were the first to describe (OSCTAP) block. They described an anatomical landmark technique and provided evidence of blockade to the mid/lower thoracic and upper lumbar spinal nerves as they travelled in the fascial plane between the transversus abdominis (TA) and internal oblique (IO) muscles.

Evidence supporting the presence of (NMDA) receptors in skin and muscles have led to the use of (MgSO4) which is NMDA antagonist via different routes.

ELIGIBILITY:
Inclusion Criteria:

* • Patients programmed for elective LC.

  * American society of anesthesiologists (ASA) physical state I or II.
  * Age over 18 years and less than 60 years old.
  * Patients of both sex are included in the study.

Exclusion Criteria:

* • Patient refusal.

  * Known hypersensitivity to the study drugs.
  * Body Mass Index > 40 kg/m2.
  * Inability to accurately describe postoperative pain to investigators.
  * Opioid tolerance or dependence.
  * Preexisting history of chronic pain.
  * History of renal, liver, cardiac, neuropsychiatric disorder problems.
  * Bleeding or coagulation abnormality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
The effect of adding different doses of MgSO4 to bupivacaine via OSCTAB block on postoperative pain according to (NRS) for 24 hours in patients scheduled for LC. | 24 hours postoperatively
  NRS Score: used to assess pain intensity . It is one of the most commonly used pain scales in medicine. The NRS consists of a numeric version of the visual analog scale. It is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible . This scale can be administered verbally. Rescue analgesia will be nalbuphine 0.1 mg/kg IV when the NRS ≥ 4.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Askar, Study Chair — Professor of Anesthesia and Intensive Care

REFERENCES:
- [Background] Grape S, Kirkham KR, Akiki L, Albrecht E. Transversus abdominis plane block versus local anesthetic wound infiltration for optimal analgesia after laparoscopic cholecystectomy: A systematic review and meta-analysis with trial sequential analysis. J Clin Anesth. 2021 Dec;75:110450. doi: 10.1016/j.jclinane.2021.110450. Epub 2021 Jul 6. PMID 34243030
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Kuscu Y, Gumus Demirbilek S. Ultrasound-guided erector spinae plane block versus oblique subcostal transversus abdominis plane block for postoperative analgesia of adult patients undergoing laparoscopic cholecystectomy: Randomized, controlled trial. J Clin Anesth. 2019 Nov;57:31-36. doi: 10.1016/j.jclinane.2019.03.012. Epub 2019 Mar 6. PMID 30851501